CLINICAL TRIAL: NCT00049881
Title: Genetic Determinants:Low HDL, High Triglycerides, Obesity
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1202; R01HL071027 (NIH)
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-01

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Hypertriglyceridemia; Obesity; Heart Diseases; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Hypertriglyceridemia; Obesity; Heart Diseases; Metabolic Syndrome

SUMMARY:
To conduct genetic studies of the metabolic syndrome characterized by very low levels of high density lipoprotein cholesterol (HDL-C), hypertriglyceridemia, and obesity.

DETAILED DESCRIPTION:
BACKGROUND:

Over the past 10 years, extensive studies have been conducted in Turkey to determine the risk factors for heart disease. Studies involving approximately 10,000 Turkish men and women from six different regions of Turkey have established that this population is unique in several ways. The Turks have the lowest plasma levels of high density lipoprotein cholesterol (HDL-C) of almost any population in the world (75 percent of the men and 50 percent of the women have HDL-C levels <40 mg/dl). The mean HDL-C levels are 10-15 mg/dl lower than those in Western European or American populations. In addition, Turks, especially Turkish women, have a tendency toward obesity [38.8 percent of the women have body mass index (BMI) >30 kg/M2], and both men and women have a tendency toward hypertriglyceridemia. The low HDL-C, however, is independent of obesity or hypertriglyceridemia. Samples from this well-characterized population provide a unique opportunity to explore the genetic determinants associated with the high prevalence of low HDL-C, hypertriglyceridemia, and obesity (characteristics of the metabolic syndrome).

The study was in response to a Request for Applications entitled "NHLBI Innovative Research Grant Program" released in July, 2001. The purpose of the initiative was to support new approaches to heart, lung, and blood diseases and sleep disorders that used existing data sets or existing biological specimen collections whether obtained through National Heart, Lung, and Blood Institute support or not.

DESIGN NARRATIVE:

The study analyzed DNA from frozen blood samples to investigate new candidate gene targets that provided insights into the abnormalities characterizing this population of Turks. The samples and extensive biodata were available on all 10,000 participants. In Specific Aim 1, the investigators identified polymorphisms in acyl CoA:diacylglycerol acyltranferase (DGAT)- I and -2 and in ATP-binding cassette A I (ABCA I) genes that were associated with differences in BMI, HDL-C, and triglyceride concentration, and other parameters such as blood pressure. These studies focussed significantly on promoter and coding sequence polymorphisms in DGAT-I and -2 and ABCAL In Specific Aim 2, the investigators determined whether the polymorphisms had functional significance by using a luciferase reporter system to determine expression of polymorphic forms of DGAT and ABCAI, a cholesterol efflux measurement to determine the functional significance of ABCAI coding sequence polymorphic sites, and a triglyceride synthesis assay to determine the functional significance of DGAT-I and -2 polymorphic sites. The polymorphic site association studies were performed on DNA samples from three subgroups of Turks: (a) individuals likely to have the metabolic syndrome, (b) individuals with isolated low HDL-C (normal triglycerides), and (c) normolipidemic unaffected controls.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mahley — J. David Gladstone Institutes